CLINICAL TRIAL: NCT01766674
Title: Specialized Centers of Research (SCOR) Kyphosis Study
Brief Title: Specialized Centers of Research (SCOR)on Sex Differences - Kyphosis Study
Acronym: SCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P0045190
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Kyphosis
Keywords: Kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kyphosis spinal exercises (Experimental): Investigator developed the intervention protocol (Kyphosis spinal exercises) of targeted spine exercises during our pilot study based upon the literature and clinical experience.We standardized the protocol with a written script and a video. Each exercise session will be preceded by light aerobic activity, ended with cool-down and stretching the neck, chest and all extremities. All participants will be carefully monitored to ensure that all exercises will be performed slowly, with correct body alignment and technique to minimize risk of injury.
  Interventions: Behavioral: Kyphosis spinal strengthening exercises
- Control (No Intervention): Control group will be enrolled in the usual care waitlist group

INTERVENTIONS:
Behavioral: Kyphosis spinal strengthening exercises — Investigator developed the intervention protocol (Kyphosis spinal exercises) of targeted spine exercises during our pilot study based upon the literature and clinical experience.We standardized the protocol with a written script and a video. Each exercise session will be preceded by light aerobic activity, ended with cool-down and stretching the neck, chest and all extremities. All participants will be carefully monitored to ensure that all exercises will be performed slowly, with correct body alignment and technique to minimize risk of injury.
  Arms: Kyphosis spinal exercises

SUMMARY:
This is a randomized, controlled trial among 100 total males and females with hyperkyphosis, aged 60 years and older, to determine the effects of an exercise intervention that includes high intensity spinal muscle strengthening exercises compared to a usual care waitlist group.

DETAILED DESCRIPTION:
Participants assigned to the intervention group will receive a high-intensity spinal strengthening group exercise program for 1 hour twice per week for 12 weeks, with home practice. The exercise program is outlined below in Table 2. The participants assigned to the control group will be receive usual care and be enrolled in a waitlist group. A physical therapist will teach the high-intensity spine strengthening exercise intervention sessions. Additionally, physical therapy graduate students will attend all exercise sessions to help ensure the safety of all participants and maintain a ratio of no more than five participants to one teacher. Participants in the control group will crossover to the spinal strengthening exercise group after 12 weeks and receive the intervention for 12 weeks.

All potential participants will be screened initially with a medical screening exam, and their primary care provider will be contacted by the study physician for approval for study participation. The participant will sign the medical release giving their primary care provider permission to release medical information to the study physician. The primary outcome will be change in Cobb angle of kyphosis over 12 weeks calculated from measurements taken from lateral spine radiographs and change in the Physical Performance Test (PPT). The investigators will also assess the effect of the exercise intervention on the secondary outcomes of physical function, strength and quality of life. The investigators will also use dual-energy x-ray absorptiometry (DXA) to determine bone mineral density before the study intervention. Study participants will receive an actigraph to measure physical activity throughout the study.

For participants in the control group who crossover to the exercise intervention group at 12 weeks will receive an additional lateral spine radiograph at the end of the intervention.

Both groups will receive a copy of the study exercise DVD at the end of the study.

Table 2. Exercise Intervention Exercises Spinal strengthening exercises (20 mins)10-12 repetitions at 70-80% 1RM Progress from 0 - 5# or theraband Spinal mobility exercises (10 mins) Passive 30 second hold Warm-up (10 mins) Increase core temperature with aerobic warm-up on bike/treadmill Prone trunk lift to neutral Spine mobilization on roller Quadruped arm/leg lift Standing shoulder flexion/thoracic extension Cool-down (5 mins) Bilateral latissimus pull-down on roller Quadruped thoracic extension mobilization Neck and upper extremity stretches Sidelying rotation and extension Spinal alignment (15 mins) Transversus abdominous strengthening Training in bilateral and single leg stance Lower extremity stretches Wall push-ups with spine in neutral Training sit-to stand, squats, lunges Diaphragmatic breathing

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* kyphosis >=40 degrees
* medical approval from primary care clinician

Exclusion Criteria:

* Gait speed <0.6 meters/sec
* inability to rise from a chair with arms crossed at chest
* painful vertebral fractures in the past 3 months
* 3 or more falls in the past year
* advanced disability or end-stage disease
* major psychiatric illness
* cognitive impairment
* alcohol, drug abuse, or narcotic pain medications
* uncontrolled hypertension
* peripheral neuropathy associated with Type I diabetes
* chest pain, myocardial infarction, or cardiac surgery within the previous 6 months
* diagnosed vestibular or neurologic disorder
* total hip or knee replacement or hip fracture within previous 6 months
* oral glucocorticoid medications for ≥ 3 months the past year
* no active movement in thoracic spine
* unable to execute exercise safety tests
* failure to comply with run-in procedures: poor attendance, or use of actigraph,
* non-English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Effect of exercise intervention on kyphosis | 3-month post baseline
  Investigators will measure change in Cobb angle on lateral spine radiograph.

SECONDARY OUTCOMES:
Effect of exercise intervention on physical function | 3-month post baseline
  Investigators will measure change in physical function with Modified Physical Performance Test (PPT), gait speed, Timed Up and Go, Timed Loaded Standing, 6 minute walk and spinal extensor muscle strength

OTHER OUTCOMES:
Effect of exercise intervention on health related quality of life (HRQOL) | 3-month post baseline
  Investigators will measure change in HRQOL with the Scoliosis Research Society SRS-30 (self image domain) and PROMIS Physical Function and Global Health Questionnaires.
Effect of exercise intervention on kyphosis | 6month post baseline for crossovers
  Investigators will measure change in Cobb angle on lateral spine radiograph
Effect of exercise intervention on physical function | 6month post baseline for crossovers
  Investigators will measure change in physical function with Modified Physical Performance Test (PPT), gait speed, Timed Up and Go, Timed Loaded Standing, 6 minute walk and spinal extensor muscle strength
Effect of exercise intervention on health related quality of life (HRQOL) | 6month post baseline for crossovers
  Investigators will measure change in HRQOL with the Scoliosis Research Society SRS-30 (self image domain) and PROMIS Physical Function and Global Health Questionnaires.
Difference in baseline characteristics and intervention effects in kyphosis in men and women | 3month post baseline
  Investigators will compare the changes in kyphosis measurements, physical function, and HRQOL in response to the intervention exercises between men and women.
Difference in baseline characteristics and intervention effects in kyphosis in men and women | 6month post baseline for crossovers
  Investigators will compare the changes in kyphosis measurements, physical function, and HRQOL in response to the intervention exercises between men and women.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Katzman, PT,DPTSc,OCS, Study Director — University of California, San Francisco; Nancy E Lane, MD, Principal Investigator — UC Davis
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Gladin A, Katzman WB, Fukuoka Y, Parimi N, Wong S, Lane NE. Secondary analysis of change in physical function after exercise intervention in older adults with hyperkyphosis and low physical function. BMC Geriatr. 2021 Feb 22;21(1):133. doi: 10.1186/s12877-021-02062-8. PMID 33618669
- [Derived] Katzman WB, Parimi N, Gladin A, Poltavskiy EA, Schafer AL, Long RK, Fan B, Wong SS, Lane NE. Sex differences in response to targeted kyphosis specific exercise and posture training in community-dwelling older adults: a randomized controlled trial. BMC Musculoskelet Disord. 2017 Dec 4;18(1):509. doi: 10.1186/s12891-017-1862-0. PMID 29202732